CLINICAL TRIAL: NCT01679067
Title: Phase IV Longitudinal Study of Gut Associated Lymphatic Tissue (GALT) in HIV (Human Immunodeficiency Virus)- Infected Patients Before and During Antiretroviral Therapy (ART)
Brief Title: Gut Associated Lymphatic Tissue (GALT) in HIV (Human Immunodeficiency Virus)- Infected Patients
Status: Completed | Type: Observational
Sponsor: Clara Lehmann (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Clara Lehmann, principal investigator, University of Cologne
Organization: University of Cologne (Other)
Other Study IDs: GALT-HIV
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: HIV Infection
Keywords: HIV; GALT
MeSH Terms: conditions — HIV Infections | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endoscopic biopsies, PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-GALT
  Interventions: Procedure: colonoscopy with endoscopic biopsies

INTERVENTIONS:
Procedure: colonoscopy with endoscopic biopsies

SUMMARY:
To date, despite the known benefits of antiretroviral therapy (ART), many HIV-infected people are presenting late with very low CD4+ T-cells levels below 350/ul. These patients are more likely to be diagnosed with opportunistic infections, their risk of death is higher and their rate of immunological improvement is slower (Mussini C et al., 2008). These patients often present a real challenge due to their advanced clinical status (Borghi V et al., 2008). Unfortunately, little is known about the clinical presentation of these patients, their responses to antiretroviral treatment and especially about the changes in the adaptive and innate immunity of the GALT.

DETAILED DESCRIPTION:
The investigator proposes to evaluate the virological, immunological and clinical outcomes of ART in HIV-1 infected 'late presenters'. The investigator further wants to investigate the longitudinal dynamics of the innate and adaptive immunity restoration in the GALT and peripheral blood of HIV infected patients under ART. In particular the investigators want to longitudinally assess DCs, NK-cells, CD4+ T-cells und CD45RO+-T-cells as well as the levels of IFNγ, IFNα, TNFα, and IL-12 in the GALT and peripheral blood by flow cytometry and by real-time PCR and correlate these data with laboratory and clinical parameters.

The investigators expect that this longitudinal study and experiments outlined in the protocol will provide valuable information about several important issues of the clinical outcome of patients under ART as well as understanding immunopathology during HIV-infection.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Patients naive to antiretroviral treatment
* Age older than 18 years
* Indication for initiation of ART
* Informed consent

Exclusion Criteria:

* Patients on antiretroviral treatment
* No informed consent
* Estimated life expectancy <1 year
* Age <18 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospective longitudinal non- controlled phase IV study, 30 patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
restoration of CD4 + T-cells in the GALT with ART | 6 months

SECONDARY OUTCOMES:
Function of Dendritic Cells (DC) in the GALT with ART | 6 months
  Functional characterization of DCs (IFNγ, IFNα) of DCs in the GALT
Functional characterization of NK-cells in the GALT with ART | 6 months
  Functional characterization on NK- cells (TNFα, and IL-12) in the GALT with ART

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cologne, Cologne, Germany